CLINICAL TRIAL: NCT04783090
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Administration Phase 1 Clinical Trial to Evalute the Satety, Tolerability, Pharmacokinetics and Preliminary Pharmacodynamics of MT1013 Injection in Healthy Subjects
Brief Title: MT1013 Clinical TRIAL In Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT1013-I-A01
Record Dates: First submitted 2021-02-20; First posted 2021-03-05 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind single-dose, sequential SAD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be double-blinded. The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (MT1013 or placebo). Blinding will be maintained until at least the clinical phase of the study is completed。
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1st cohort (Experimental): MT1013 injection at 2.5 mg.
  Interventions: Drug: MT1013
- 2nd cohort (Experimental): MT1013 injection at 5 mg.
  Interventions: Drug: MT1013
- 3rd cohort (Experimental): MT1013 injection at 10 mg.
  Interventions: Drug: MT1013
- 4th cohort (Experimental): MT1013 injection at 15 mg.
  Interventions: Drug: MT1013
- 5th cohort (Experimental): MT1013 injection at 20 mg.
  Interventions: Drug: MT1013

INTERVENTIONS:
Drug: MT1013 — bispecific peptide as a CaSR agonist and a functional OGP analogue

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose administration phase one clinical trial to evaluate the safety, tolerability, pharmacokinetics and preliminary pharmacodynamics of MT1013 injection in healthy subjects.

DETAILED DESCRIPTION:
This will be a single center, Phase 1, randomized, double-blind single-dose, sequential SAD study.

This SAD study will consist of up to 5 cohorts (1 cohort per dose level). Each cohort will include 8 subjects (6 subjects receiving the active study drug and 2 subjects receiving matching placebo).

A staggered dosing schedule will be used for each dose level administered under fasting conditions. Two (2) sentinel subjects (1 active and 1 placebo) will be dosed first (a minimum of 1 hour apart) and the remaining 6 subjects will be dosed no sooner than the next day (each dosed at least 15 minutes apart).

Following completion of each dose level, a SRC will review the safety and tolerability data as well as the available PK data up to 48 hours in order to make decisions whether to escalate to the next dose level, decrease the next dose level, repeat a dose level, or to not evaluate any additional dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤55 years of age, with BMI >18.0 and <30.0 kg/m2 and body weight ≥45.0 kg for males and females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, GI, renal, hepatic, and metabolic disease.
3. Females of childbearing potential who are sexually active with a non-sterile male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:
4. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, hepatitis C, or Treponema pallidum antibody found during medical screening.
2. Positive urine drug screen or urine cotinine test or alcohol breath test at screening.
3. Positive fecal occult blood test at screening.
4. History of clinically significant drug allergies.
5. Positive pregnancy test at screening.
6. Clinically significant ECG abnormalities (QTcF ≥450 ms) or a family history of long QT syndrome.
7. Clinically significant vital sign abnormalities at screening.
8. History of significant alcohol abuse within 1 year prior to screening.
9. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
10. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days or 5 half-lives (whichever is longer) prior to the first dosing.
11. Use of prohibited medications for the timeframes specified.
12. Donation of plasma within 7 days prior to dosing.
13. Breast-feeding subject.
14. The combination of diseases that may affect the assessment of drug absorption, distribution, metabolism, excretion and safety data, or that can reduce compliance.
15. Subjects with previous clinically significant history of epileptic seizures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MT1013 for injection in healthy adult subjects. | Three months
  Assessment of adverse events

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of MT1013 for injection in healthy adult subjects | 3 days
  AUC0-t
PK | 3 days
  AUC0-inf
PK | 3 days
  Cmax
PK | 3 days
  Tmax
PK | 3 days
  T½ el
To characterize the pharmacodynamics (PD) of MT1013 for injection in healthy adult subjects | 3 days
  Serum PTH value
PD | 3 days
  Serum total calcium value
PD | 3 days
  serum phosphorous value

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No